CLINICAL TRIAL: NCT01249859
Title: Has the Quota of Signet Ring Cells an Influence on Prognosis and Treatment Strategy in the Upper GI Tract Adenocarcinomas?
Brief Title: Prognosis of Signet Ring Cells in Upper Digestive Neoplasms
Acronym: ADCI001
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: ADCI 001
Record Dates: First submitted 2010-10-26; First posted 2010-11-30 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Signet Ring Cell Carcinoma; Stomach Disease; Oesophagus; Prognostic; Case-control Study
Keywords: stomach disease; signet ring cell carcinoma; chemotherapy; Prognostic
MeSH Terms: conditions — Carcinoma, Signet Ring Cell; Stomach Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Signet ring cell carcinoma
- non signet ring cell adenocarcinoma

SUMMARY:
Background • A major increase in incidence of signet ring cell adenocarcinomas (ADCI) of the upper digestive tract in western countries

* Discordant results in the literature concerning the prognosis value of the presence of signet ring cells.
* Preliminary data suggesting (i) an advanced stage at time of diagnosis, (ii) more often in the form of carcinose, (iii) a more pejorative prognosis, (iv) a recurrence more frequent, more quickly, and more often in the form of peritoneal carcinose, (v) a chemo resistance (vi) the need for a specific therapeutic strategy compared to non-signet ring cell adenocarcinomas.

Primary objective To test the hypothesis that 5-year survival rate is significantly lower in the signet ring cells (SRC) adenocarcinoma when compared to non-SRC adenocarcinoma in the upper digestive tract

Secondary objectives

* Impact of neoadjuvant CT on overall survival
* Impact and differential diagnostic value of linitis
* R0 resection rates
* 3 years recurrence free survival
* Overall 3 years survival
* Prognostic factors
* Prognostic value of the presence of a minority quota of signet ring cell
* Objective response rate after medical treatment (chemotherapy, radiochemotherapy) in non-resected patients
* Tolerance of (radio) chemotherapy for ADCI

Methodology Intention to treat retrospective case-control multicentric study A pairing on demographic criteria (age, sex, ASA score, center) and tumor criteria (TNM stage) will be done to ensure comparability in case control study groups.

Inclusion criteria All consecutive patients taken care of, for a proven histologically adenocarcinoma (ADCI and ADNCI) of the esophagus, the esogastric junction, or the stomach, in surgical or medical oncology investigator centers, will be saved in a given database.

For whom the first consultation took place between January 1997 and January 2010

Exclusion criteria Histological type other than adenocarcinoma Other localization than esogastric junction, esophagus or stomach

Planned study period The data will be collected over a period from January 1997 to January 2010.

The objective is to complete the data collection for summer 2010.

DETAILED DESCRIPTION:
stomach cancer signet ring cell carcinoma prognosis chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients taken care of, for a proven histologically adenocarcinoma (ADCI and ADNCI) of the esophagus, the esogastric junction, or the stomach, in surgical or medical oncology investigator centers, will be saved in a given database.
* For whom the first consultation took place between January 1997 and January 2010
* As they benefit from a medical and/or surgical support (primitive cancer being or not resected), whatever the metastatic or the recurrence situation was.

Exclusion Criteria:

* Histological type other than adenocarcinoma
* Other localization than esogastric junction, esophagus or stomach

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intention to treat retrospective case control multicentric study, Patients will be divided into two groups (ADCI or ADNCI) depending on the presence or not of signet ring cells on definitive histologic analysis Another analysis based on chemo administration or not will be provided A pairing on demographic criteria (age, sex, ASA score, center, TNM stage and will be done to ensure comparability in case control study groups.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that 5-year survival rate is significantly lower in the signet ring cells (SRC) adenocarcinoma when compared to non-SRC adenocarcinoma in the upper digestive tract | participants are followed until death or time point at 31 september 2010

SECONDARY OUTCOMES:
3 year recurrence free survival | participants are followed until recurrence or time point at 31 september 2010
Overall 3 year survival according to tumor stage, node invasion, and tumor localization | participants are followed until death or time point at 31 september 2010

CONTACTS AND LOCATIONS:
Overall Officials: christophe mariette, MD, PhD, Study Director — CHU lille
Locations (1):
- University Hospital of Lille, Lille, France

REFERENCES:
- [Derived] Robb WB, Messager M, Goere D, Pichot-Delahaye V, Lefevre JH, Louis D, Guiramand J, Kraft K, Mariette C; FREGATWorking Group-FRENCH. Predictive factors of postoperative mortality after junctional and gastric adenocarcinoma resection. JAMA Surg. 2013 Jul;148(7):624-31. doi: 10.1001/jamasurg.2013.63. PMID 23552982
- [Derived] Messager M, Lefevre JH, Pichot-Delahaye V, Souadka A, Piessen G, Mariette C; FREGAT working group - FRENCH. The impact of perioperative chemotherapy on survival in patients with gastric signet ring cell adenocarcinoma: a multicenter comparative study. Ann Surg. 2011 Nov;254(5):684-93; discussion 693. doi: 10.1097/SLA.0b013e3182352647. PMID 22005144